CLINICAL TRIAL: NCT05887076
Title: Postoperative Delirium After Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anaesthesiology and Intensive Care Medicine CCM/CVK, Charite University, Berlin, Germany
Other Study IDs: PODNTX
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Post-operative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a retrospective evaluation of the routine data of patients who underwent a kidney transplant at the Charité Campus Mitte between January 2015 and December 2019 (until the corona pandemic).

DETAILED DESCRIPTION:
Post-anesthetic complications such as delirium can occur in patients after kidney transplantation. We would therefore like to characterize pathophysiological changes after transplantation of the kidneys and, if necessary, gain diagnostic and therapeutic knowledge. The purpose is to study postoperative delirium after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older who underwent kidney transplantation and who were admitted to Post-intensive care unit or to an Intensive care unit at the Campus Charité Mitte

Exclusion Criteria:

* Incomplete data records of the parameters to be determined
* Underage Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients 18 years and older who underwent kidney transplantation
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | 2015 - 2019
  Incidence of delirium is recorded from validated delirium scores.

SECONDARY OUTCOMES:
Duration of delirium | 2015 - 2019
  Duration of delirium is recorded in days.
Severity of delirium | 2015 - 2019
  Severity of delirium is recorded from validated delirium scores.
Intraoperative parameter | 2015 - 2019
  Intraoperative parameter are recorded from patients with delirium.
Anesthesia | 2015 - 2019
  Anesthesia is recorded from patient files of patients with delirium.
Anesthesiological parameters | 2015 - 2019
  Anesthesiological parameters are recorded from patient files of patients with delirium.
Immunosupressive therapy | 2015 - 2019
  Immunosupressive therapy is recorded in patients with delirium.
Delirium treatment | 2015 - 2019
  Delirium treatment is recorded peri-operatively.
Pain teatment | 2015 - 2019
  Pain treatment is recorded peri-operatively.
Intensive care unit stay | 2015 - 2019
  Length of intensive care unit stay is measured in days.
Hospital stay | 2015 - 2019
  Length of hospital stay is measured in days.
Mortality | 2015 - 2019
  Mortality is measured within the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Anaesthesiology and Intensive Care Medicine CCM, Charite - Universitätsmedizin, Berlin
  - Medical Clinic with a focus on Nephrology and Internal Intensive Care Medicine, Berlin

IPD SHARING:
Plan to Share IPD: No